CLINICAL TRIAL: NCT06203535
Title: Effect of Aerobic Training on Quality of Life in Elderly With Idiopathic Chronic Fatigue
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pharos University in Alexandria (Other)
Responsible Party: Principal Investigator, Ola Mohamed Elsayed Elgohary, lecturer of physical therapy pharos university, Pharos University in Alexandria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aerobic training and fatigue
Record Dates: First submitted 2023-12-11; First posted 2024-01-12 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-12

CONDITIONS: Chronic Idiopathic Fatigue
Keywords: aerobic training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic training (group a) (Experimental): In addition to the standard physical therapy exercise programme (which includes flexibility and balance exercises), twenty individuals with idiopathic chronic fatigue will participate in an aerobic training group and walk for 45 minutes on a treadmill three times a week for two months. The workouts began with a five- to ten-minute warm-up on the treadmill and concluded with an equally extended cool-down. Using the Karvonen method, for exercise intensities ranging from 60 to 75 per cent of heart rate reserve during a 35-minute group cumulative exercise session.
  Interventions: Other: Aerobic training
- control group (group B) (Experimental): twenty participants have idiopathic chronic fatigue will received only traditional physical therapy exercise program (flexibility and balance activities)
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Aerobic training — In addition to the standard physical therapy exercise programme (which includes flexibility and balance exercises), twenty individuals with idiopathic chronic fatigue will participate in an aerobic training group and walk for 45 minutes on a treadmill three times a week for two months. The workouts began with a five- to ten-minute warm-up on the treadmill and concluded with an equally extended cool-down. Using the Karvonen method, for exercise intensities range from 60 to 75 percent of heart rate reserve during a 35-minute group cumulative exercise session.
  Other Names: traditional physical therapy exersise program

SUMMARY:
the study was conducted to evaluate the effectiveness of aerobic training for decreasing fatigue severity and increasing quality of life in elderly with idiopathic chronic

DETAILED DESCRIPTION:
idiopathic chronic fatigue (ICF) or chronic idiopathic fatigue (CIF), this type of tiredness is ongoing and unrelated to any underlying medical or mental health issues. Different diagnostic criteria apply to people with idiopathic chronic fatigue and those with chronic fatigue syndrome (CFS).

Regular aerobic exercise has been demonstrated to improve cardiopulmonary fitness, increase physical activity levels, and decrease the degree of fatigue in elderly patients with severe idiopathic fatigue.

ELIGIBILITY:
inclusion criteria:

* ages ranged from 60 to 70 years and they will have BMI in between25.0-29.9 kg/m2,
* complaining fatigue least six months ago without identifying any specific cause for their fatigue.
* could walk safely without the aid of another person.

Exclusion Criteria:

* Renal, vascular, hepatic, autoimmune, heart, chest and thyroid disorders.
* Lower limb arthritis or any orthopedic problem will hinder the training.
* Cognitive impairment or psychological problems,
* fatigue caused as a known side effect of medication.
* any febrile condition and/or infectious diseases

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-04-13 (Estimated); Study Completion 2024-05-07 (Estimated)

PRIMARY OUTCOMES:
Older People's Quality of Life Questionnaire (OPQOL-brief): | 2 monthes will take pre and post total study peroid
  Thirteen items make up the questionnaire; one item includes codes of Strongly agree (1), Agree (2), Neither (3), Disagree (4), and Strongly disagree (5). Positive items are reverse coded to indicate higher quality of life (QoL) with higher scores once all of the questions have been added up to give an overall OPQOL-Brief score.
fatigue severity assessment scale | 2 month will take pre and post total study peroid
  Before and during the study period, the physical and mental weariness of both groups (A and B) was measured using a straightforward ten-item fatigue scale. The participants rated an etch statement from five categories, from never to always, using a scale. 1 denotes never, 2 occasionally, 3 regularly, 4 often and 5 always worn out. The greater figure denotes an extremely high degree of exhaustion and fatigue.
six mints walk test | 2 monthes will take pre and post total study peroid
  Before and during the study period, the aerobic capacity and endurance of both groups (A and B) were assessed using this sub-maximal test. The outcomes were compared to see how the performance capacity changed with walks lasting longer than six minutes.
Glutathione blood test: | 2 monthes will take pre and post total study peroid
  Glutathione is an antioxidant, a type of chemical which helps to boost the immune system as well as prevent and reverse cellular damage. Glutathione levels tend to decrease naturally with age as well as due to health conditions such as liver disease, insomnia, and chronic disease.Before and after the study period, venous blood was taken from both groups (A and B) at baseline when they were not fasting. Tandem mass spectroscopy was used to analyse the samples and determine the degree of serum changes in both study groups based on their respective treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen FT, Etnier JL, Chan KH, Chiu PK, Hung TM, Chang YK. Effects of Exercise Training Interventions on Executive Function in Older Adults: A Systematic Review and Meta-Analysis. Sports Med. 2020 Aug;50(8):1451-1467. doi: 10.1007/s40279-020-01292-x. PMID 32447717
- [Background] Hendriks C, Drent M, Elfferich M, De Vries J. The Fatigue Assessment Scale: quality and availability in sarcoidosis and other diseases. Curr Opin Pulm Med. 2018 Sep;24(5):495-503. doi: 10.1097/MCP.0000000000000496. PMID 29889115
- [Background] Bowling A, Hankins M, Windle G, Bilotta C, Grant R. A short measure of quality of life in older age: the performance of the brief Older People's Quality of Life questionnaire (OPQOL-brief). Arch Gerontol Geriatr. 2013 Jan-Feb;56(1):181-7. doi: 10.1016/j.archger.2012.08.012. Epub 2012 Sep 19. PMID 22999305